CLINICAL TRIAL: NCT00375778
Title: Parkinson's Disease Evaluated by Positron Emission Tomography and the Effect of the NMDA Receptor Antagonist Memantine
Brief Title: Parkinson's Disease Evaluated by PET and the Effect of Memantine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-004139-74
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Positron Emission Tomography; Memantine; NMDA antagonists; Cerebral Blood Flow; Cerebral Metabolic Rate of Oxygen
MeSH Terms: conditions — Parkinson Disease | interventions — Memantine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: memantine (drug)

SUMMARY:
Purpose of study: To investigate whether the NMDA antagonist Memantine has a substantial effect of brain metabolism in patients with Parkinson's disease (PD), using Positron Emission Tomography (PET).

Background: Disturbances in brain metabolism is thought to contribute to degeneration of neurons in brain of PD patients. Production of toxic oxygen radicals and presence of too much excitatory neurotransmitter (glutamate) due to over activity is involved. These factors can theoretically be alleviated by memantine.

Hypothesis: Memantine decreases metabolism in areas in PD brain known to be over-active. Decreases in cerebral blood flow and oxygen metabolism in these areas will be the consequence and this can be detected by PET.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease (British Brain Bank Criteria)
* Age 50-70y

Exclusion Criteria:

* Tobacco use
* Any serious medical conditions (Heart disease, kidney disease, liver disease, endocrinological disorders etc)
* Metal implants contraindicating MR scan
* Drug use affecting the central nervous system
* Psychiatric disorders
* Head trauma or any disorders of the head, skull or brain
* Drug addiction or use of any kind of illegal substance affecting the central nervous system
* Pregnancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-04; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ostergaard, MD, Ph.D, Principal Investigator — Aarhus University Hospital
Locations (1):
- PET center, Aarhus University Hospital, Aarhus, Denmark